CLINICAL TRIAL: NCT00218101
Title: Dose Reduction Strategies in Oral Opioid Dependence Subsequent to Pain Management: An Exploratory Study
Brief Title: Buprenorphine as a Treatment for Individuals Dependent on Analgesic Opioids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Texas (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-09262-11; P50-09262-11; DPMC
Record Dates: First submitted 2005-09-16; First posted 2005-09-22 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-10

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
Opioids used to treat chronic pain have a high abuse potential. The purpose of this study is to determine the effectiveness of buprenorphine in treating opioid dependent individuals who abuse opioids that are prescribed for chronic pain.

DETAILED DESCRIPTION:
Many individuals who take opioids for chronic pain abuse the opioid medication. Buprenorphine is an opioid partial agonist that may be effective in treating individuals who abuse opiate pain medication. The purpose of this study is to compare two buprenorphine dosing regimens in order to determine which regimen is more effective in reducing opiate pain medication use and facilitating successful opioid detoxification.

This study will last 27 weeks. Participants will receive a maintenance dose of 8 mg of buprenorphine for 6 weeks, followed by a dose reduction in 2 mg increments over the course of the following 20 weeks. All participants will attend weekly clinical management sessions for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Current opioid analgesic dependence
* History of at least 2 years of oral opiate analgesic use
* Prescribed opioids for chronic pain
* Pain episode of at least 6 months duration within the 5 years prior to study entry
* Available for the duration of the study
* Good general health

Exclusion Criteria:

* Currently using any illicit substance
* Meets criteria for alcohol dependence
* History of heroin use
* History of opiate replacement therapy, including Levo-Alpha Acetyl Methadol (LAAM) or methadone
* Evidence of current maximal primary pain

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10
Dates: Start 2004-05; Study Completion 2005-03

PRIMARY OUTCOMES:
Substance use
medication compliance
treatment retention

SECONDARY OUTCOMES:
Behavioral and psychological measures (measured during the dose reduction phase)

CONTACTS AND LOCATIONS:
Overall Officials: John Grabowski, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Health Science Center, Houston, Texas, United States